CLINICAL TRIAL: NCT02470793
Title: Technique And Results Evaluation In Endothelial Keratoplasty
Brief Title: Technique And Results In Endothelial Keratoplasty
Acronym: TREK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EDUARD PEDEMONTE-SARRIAS (Other)
Responsible Party: Sponsor-Investigator, EDUARD PEDEMONTE-SARRIAS, MEDICAL DOCTOR, Hospital Mutua de Terrassa
Organization: Hospital Mutua de Terrassa (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00001
Record Dates: First submitted 2015-06-06; First posted 2015-06-12 (Estimated); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Corneal Endothelial Cell Loss; Fuchs' Endothelial Dystrophy
Keywords: Corneal Endothelial Cell Loss; Fuchs' Endothelial Dystrophy; Lamellar Keratoplasty; Descemet Stripping Endothelial Keratoplasty; Descemet Membrane Endothelial Keratoplasty; Minimal Surgical Procedure
MeSH Terms: conditions — Corneal Endothelial Cell Loss; Fuchs' Endothelial Dystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DSAEK group (Active Comparator): Subjects operated of Descemet Stripping Automated Endothelial Keratoplasty.
  Interventions: Procedure: Descemet Stripping Automated Endothelial Keratoplasty
- DMEK group (Experimental): Subjects operated of Descemet Membrane Endothelial Keratoplasty.
  Interventions: Procedure: Descemet Membrane Endothelial Keratoplasty

INTERVENTIONS:
Procedure: Descemet Stripping Automated Endothelial Keratoplasty — Descemet Stripping Automated Endothelial Keratoplasty
  Other Names: DSAEK; DSEK
  Arms: DSAEK group
Procedure: Descemet Membrane Endothelial Keratoplasty — Descemet Membrane Endothelial Keratoplasty
  Other Names: DMEK
  Arms: DMEK group

SUMMARY:
To assess and compare the complications and results of different lamellar endothelial keratoplasty techniques and its variations.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis with corneal endothelial dysfunction requiring lamellar endothelial corneal transplantation.
2. Free acceptance to be enrolled in the trial, and signature of the informed consent by the subject and/or its legal representatives.

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Visual acuity | First six months postoperatively

SECONDARY OUTCOMES:
Endothelial cell density | First six months postoperatively
Intraoperative complications | First six months postoperatively
Postoperative complications | First six months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Eduard Pedemonte-Sarrias, MD, Principal Investigator — Hospital Universitari Mútua Terrassa
Locations (1):
- Hospital Universitari Mutua Terrassa, Terrassa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided